CLINICAL TRIAL: NCT04441593
Title: Internet-based Videoconferencing to Address Alcohol Use and Pain Among People With HIV
Brief Title: Internet-based Video-conferencing to Address Alcohol Use and Pain: a Pilot Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4546 [Study 3]; UH3AA026192 (NIH)
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Alcohol Drinking and Chronic Pain Intervention; Control Condition
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol; Methods; Therapeutics

STUDY DESIGN:
Intervention Model Description: Compare Intervention to Control Condition in a Between Subjects Design
Who Masked: Outcomes Assessor
Masking Description: Three and six month assessments will be conducted by RA who is masked to intervention condition
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Videoconferencing Intervention for Heavy Drinking and Chronic Pain
  Interventions: Behavioral: Motivational and Cognitive-Behavioral Management for Alcohol and Pain (MCBMAP)
- Control (Active Comparator): Treatment as Usual
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Motivational and Cognitive-Behavioral Management for Alcohol and Pain (MCBMAP) — Videoconferencing intervention to reduce alcohol use and chronic pain interference and severity
  Other Names: Intervention
  Arms: Intervention
Behavioral: Treatment as Usual — Psychoeducation and Information about Treatment Resources
  Other Names: Control
  Arms: Control

SUMMARY:
This pilot study seeks to provide effect size estimates and test feasibility of a novel, integrated behavioral approach to reduce heavy drinking and chronic pain among patients in HIV-care delivered via internet-based videoconferencing.

DETAILED DESCRIPTION:
This pilot study is a between-groups design to compare a novel integrated behavioral video telehealth intervention for heavy drinking PLWH with chronic pain to a control condition. Forty-eight heavy drinking patients in HIV-care with moderate or greater pain will be recruited for the study. Following baseline assessment, participants will be randomly assigned to either intervention or control conditions. Participants will complete assessment measures of heavy drinking and pain interference/severity at 3 and 6 months post-baseline. Secondary alcohol outcomes will include alcohol-related consequences

ELIGIBILITY:
Inclusion Criteria:

* engaged in HIV care, heavy drinking defined as more than 7/14 drinks per week for women/men or by a single episode of 4/5 (women/men), chronic (at least 3 months duration) moderate or greater (4 or more on the severity scale of the BPI, and non-cancer related pain

Exclusion Criteria:

* psychoactive medication for pain or alcohol use for fewer than 2 months
* history of bipolar disorder or schizophrenia
* current expressed suicidal intent
* prior history of alcohol withdrawal related seizures or delirium tremens
* current behavioral treatment for pain or alcohol use
* any scheduled surgery within the next 6 months or acute life threatening illness that requires treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
Alcohol Time Line Follow-Back (30)- Heavy Drinking Episodes | Past 30 days
  Number of heavy drinking episodes NIAAA criteria (5+drinks men/ 4+ drinks women)
Alcohol Time Line Follow-Back (30) - Average Drinks per Week | Past 30 days
  Average number of standard alcohol-containing drinks in the past 30 days
Brief Pain Inventory - Pain Severity | Past 7 days
  BPI is an 11-point scale anchored with "0" best and "10" is worst Scale range 0-10
Brief Pain Inventory - Pain Interference | Past 7-Days
  BPI is an 11-point scale anchored with "0" best and "10" is worst Scale range 0-10. Pain Interference is measured as the mean of 7-items each rated on an 11-point scale

SECONDARY OUTCOMES:
Short Inventory of Alcohol Problems-Revised | 3 months
  17-item measure with 4-point Likert scale items ranging from "0" never to "3" daily/almost daily. Scale range 0-51
Goal Systems Assessment Battery-Alcohol | Past 30 days
  Ratings of self-regulatory capacities related to reducing alcohol use. Items are 5-point Likert-scales. There are 4 subscales utilized including planning, monitoring, self-efficacy, and value. Higher scores indicate better outcomes
Goal Systems Assessment Battery-Pain | Past 30 days
  Ratings of self-regulatory capacities related to reducing alcohol use. Items are 5-point Likert-scales. There are 4 subscales utilized including planning, monitoring, self-efficacy, and value. Higher scores indicate better outcomes

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Boston University Department of Psychological and Brain Sciences, Boston, Massachusetts
  - General Clinical Research Unit, Boston University, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
For proposals that contain analyses that are not already planned or in progress, the investigators will make data available for collaboration with a study investigator, provided IRB and other appropriate regulatory approvals are obtained (including but not limited to Federal and Boston University IRB review and approval). Data to be shared will be de-identified to minimize the risk of deductive disclosure. Documentation will be provided for all shared data including copies of data collection forms, schedule of study assessments, data dictionaries documenting all original and derived variables, descriptive statistics for all variables included in the data sets, and a written description of the study conduct and noteworthy details anticipated to potentially affect data interpretation. Costs associated with producing data sets and analysis will be the responsibility of investigators seeking the data.
Supporting Information: Study Protocol, ICF
Time Frame: Twelve months following request, de-identified data will be available to investigators upon request. This access will be provided for 7 years following publication of main trial
Access Criteria: Specific data may be shared based on proposals received and reviewed by the study investigators and determined to have scientific merit. Limited public-use data sets may also be prepared and made available in a web-data archive to be developed and maintained by the data coordinating center (BEDAC).